CLINICAL TRIAL: NCT02366936
Title: Effectiveness of Tortle Midliner Positioning System on the Prevention and Treatment of Cranial Molding Deformities in Preterm Infants
Brief Title: Treatment of Cranial Molding Deformities in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Tortle Products LLC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00060408
Record Dates: First submitted 2015-02-12; First posted 2015-02-19 (Estimated); Results first posted 2017-04-18 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2017-03

CONDITIONS: Preterm Infants; Dolichocephaly; Positional Scaphocephaly

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Use of Tortle midliner (Experimental): This study will be an interventional, longitudinal study of 30 preterm infants using the Tortle Midliner.
  Interventions: Device: Tortle Midliner

INTERVENTIONS:
Device: Tortle Midliner — The Tortle Midliner is a breathable, knit beanie with two support rolls to help position the infant's head in midline while supine. It can also be worn sidelying or prone. The design includes Velcro adjustments and tabs for nasal cannula and feeding tubes. It is compatible with some ventilation devices, nasal CPAP, X-ray, and bilirubin shades. The beanie is designed to prevent dolichocephaly and provide passive stretch to cervical rotators if head preference has developed. It comes in three sizes and can fit preemies weighing 500 to 2500 g.

SUMMARY:
The purpose of this study is to determine the effectiveness of the Tortle Midliner positioning system in prevention and/or treatment of dolichocephaly, which can develop in preterm infants during the hospital stay.

Specific Aim: Determine if the use of the Tortle Midliner is a more effective prevention and treatment strategy for dolichocephaly than current standard of care intervention in the Duke Intensive Care Nursery (ICN).

DETAILED DESCRIPTION:
Dolichocephaly (or positional scaphocephaly) is defined as a boat-shaped or elongated anterior-posterior axis as a result of skull flattening during side-to-side head positioning of infants during hospitalization. This deformity often takes place in preterm infants <32 weeks because the preferred position is sidelying or prone for improved ease of containment, decreased reflux episodes, and decreased apnea/bradycardia. Supine positioning with head in midline is recommended to decrease the occurrence of this deformity, but maintaining midline is difficult as a result of gravity and preterm hypotonia. Developmental positioning through use of special positioning aids and caregiver education are common interventions used to address dolichocephaly. Dolichocephaly may resolve prior to hospital discharge, but in some cases infants are discharged home with the deformity.

Despite documentation of dolichocephaly in preterm infants for nearly three decades, few studies report how often it occurs or the rate of resolution with intervention. Prematurity appears to be the most common predetermining factor. Preterm infants may experience a limited variety of positions due to autonomic instability or critical respiratory status. These infants are often positioned in prone to improve oxygenation and decrease incidence of reflux. Furthermore, the preterm infant demonstrates proximal hypotonia, causing the head to fall to either side with gravity while in supine. Bilateral flattening of the lateral skull develops as a result of the weight of the head and the pressure of gravity.

The correlation between low birth weight and head flattening has been established in the literature. Researchers suggested that the deformity was preventable with the use of air or water pillows. Limited emphasis was placed on body position (i.e. supine, sidelying, or prone) in these articles. Since this period of time, the use of positioning aids and developmental positioning has been used to decrease the occurrence of dolichocephaly during hospitalization. Despite these interventions, some infants have dolichocephaly at hospital discharge.

The long-term consequences of dolichocephaly are not fully known, but it has been correlated with delayed reaching skills, tightness in the spinal extensors and scapular retractors, and development of motor asymmetries. Other long-term effects of dolichocephaly have been evaluated minimally. Elliman's study demonstrated comparable developmental quotients at age 3 when comparing a preterm group to controls. Kitchen and colleagues reported no differences in IQ at a 7-year follow up. Mewes and colleagues, however, suggest that the shift in cortical structures, caused by dolichocephaly may affect the preterm brain, which continues to develop rapidly after birth. Since the American Academy of Pediatrics established the widely successful and influential "Back to Sleep Campaign" in 1992, many studies have established the relationship between prevalence and long-term neuro-developmental outcomes of preterm infants with plagiocephaly - asymmetric flattening of the skull due to head preference - but there are no studies that determine the long-term neuro-developmental outcomes of preterm infants with dolichocephaly. Increased time spent supine, coupled with the fact that nearly half of preterm infants leave the hospital with a head preference, calls for updated long-term study of the effect of dolichocephaly specifically on neuro-developmental outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Birth weight of <1500 g
2. Gestational age of ≤ 30 weeks
3. <2 weeks chronological age
4. ≤30 weeks gestation at time of parent consent
5. Receiving continuous positive airway pressure (CPAP), nasal cannula or room air
6. Signed the informed consent from the legal caregiver

Exclusion Criteria:

1. Determined to be too medically unstable by their attending physician
2. Diagnosed with a genetic/chromosomal abnormality, congenital neuromuscular disorder, craniofacial abnormalities, congenital hydrocephalus, post-hemorrhagic hydrocephalus, or other diagnoses determined by the PI that impacts generalizability of results

Ages: 23 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2015-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Malcolm, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Use of Tortle Midliner
Started | 32
Completed | 24
Not Completed | 8
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 4
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Use of Tortle Midliner
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 32
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 23
  White | 8
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 32
Gestational age [Mean (Full Range); unit: weeks] | 27 [25 to 30]
Birth weight [Mean (Full Range); unit: g] | 975 [590 to 1430]

OUTCOME MEASURES:

1. Primary Outcome: Cranial Index (CI)
Description: CI was determined by calculating the ratio of the biparietal diameter (BiPD) over the occipitofrontal diameter (OFD). The BiPD is defined as the widest transverse diameter of the head. BiPD was measured from the most prominent lateral point on each side of the skull in the area of parietal and temporal bones. The OFD is defined as the diameter of the head from the most prominent midline point of the frontal bone (glabella) to the occipital protuberance. While various reported ranges exist for cranial molding norms, dolichocephaly was defined as a CI of <76%. The normative CI range is 76-85% for prone and supine sleeping infants.
  CI = BPD/OFD x 100
Time Frame: 34 weeks gestational age
Measure: Median (Full Range); unit: cranial index
Arm/Group | Use of Tortle Midliner
Number analyzed (Participants) | 24
cranial index | 79 [73 to 83]

2. Primary Outcome: Number of Infants That Developed Dolichocephaly by the End of the Study
Description: dolichocephaly for this study is considered a cranial Index <76% at 34 weeks post menstrual age (PMA)
Time Frame: 34 weeks gestational age
Measure: Number; unit: participants
Arm/Group | Use of Tortle Midliner
Number analyzed (Participants) | 24
participants | 3

ADVERSE EVENTS:
Time Frame: 1year, 3 months
Arm/Group | Use of Tortle Midliner
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 1/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Use of Tortle Midliner (N=32)
non-blanchable pressure ulcer (Investigations) | 1

LIMITATIONS AND CAVEATS:
Study used the original design of the Tortle Midliner (TM). TM's new design adjustments (multiple velcro attachments, material to prevent slippage inside the cap, and doesn't cover head) may result in different outcomes based on our study protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes